CLINICAL TRIAL: NCT03735628
Title: An Open-label, Multi-center, Phase 1b/2 Study to Evaluate the Safety and Efficacy of Copanlisib in Combination With Nivolumab in Patients With Advanced Solid Tumors.
Brief Title: An Study to Evaluate the Safety and Efficacy of Copanlisib in Combination With Nivolumab in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19769
Record Dates: First submitted 2018-10-25; First posted 2018-11-08 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Non-small Cell Lung Cancer (NSCLC); Head and Neck Squamous Cell Carcinoma (HNSCC); Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Hepatocellular | interventions — copanlisib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose escalation (Experimental): Copanlisib:
  45 mg (dose level -1) or 60 mg (dose level 1) on Day 1, Day 8 and Day 15 (28 day cycle)
  Nivolumab:
  240 mg on Day 15 of Cycle 1 and on Day 1 and Day 15 of subsequent cycles (28 day cycle).
  Interventions: Drug: Copanlisib; Drug: Nivolumab
- Dose expansion (Experimental): Copanlisib:
  Recommended phase 2 dose established in the phase 1b part on Day 1, Day 8 and Day 15 (28 day cycle)
  Nivolumab:
  240 mg on Day 15 of Cycle 1 and on Day 1 and Day 15 of subsequent cycles (28 day cycle).
  Interventions: Drug: Copanlisib; Drug: Nivolumab

INTERVENTIONS:
Drug: Copanlisib — Copanlisib: lyophilisate for reconstitution and further dilution for infusion
Drug: Nivolumab — Nivolumab: concentrate for solution for infusion

SUMMARY:
The purpose of the dose escalation part of this study is to determine the feasibility of using the combination of copanlisib and nivolumab in subjects with advanced solid tumors, and to determine the maximum tolerated dose of copanlisib in combination with nivolumab. The maximum tolerated dose will then be used in Phase 2 (dose expansion) of the study.

DETAILED DESCRIPTION:
Study was originally designed with both Phase I and Phase II part, but sponsor decided not to conduct Phase 2 part due to strategic portfolio re-prioritization.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a histologically confirmed diagnosis of:

Phase 1b:

* Advanced solid tumors where nivolumab is indicated as per the latest nivolumab Prescribing Information,

Phase 2:

* Metastatic NSCLC, progressing on or after prior pembrolizumab therapy with or without chemotherapy, irrespective of PD-L1 expression Patients with EGFR or ALK genomic tumor aberrations should have disease progression on FDA-approved therapy for these aberrations.
* Recurrent or metastatic HNSCC progressing on or after prior pembrolizumab therapy with or without chemotherapy
* HCC progressing after any prior therapy.

Exclusion Criteria:

* Active, known or suspected autoimmune disease. Participants with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Major surgery, open biopsy or significant traumatic injury ≤ 28 days prior to first administration of study intervention. Central line surgery is not considered major surgery
* Symptomatic metastatic brain or meningeal carcinomatosis or tumors unless the participant is > 6 months from definitive therapy (surgery or radiotherapy), has no evidence of tumor growth on an imaging study and is clinically stable with respect to the tumor at the start of study intervention.
* Other malignancy within the last 5 years except for the following, which are permitted:

  * curatively treated basal cell/squamous cell skin cancer,
  * carcinoma in situ of the cervix,
  * superficial transitional cell bladder carcinoma (if BCG [Bacillus Calmette-Guerin] treatment was given, there should be a minimum of 6 months between last dose and enrollment),
  * in situ ductal carcinoma of the breast after complete resection,
  * participants with localized, resected and/or low-risk prostate cancer may be eligible after discussion with the sponsor's designated medical representative and sponsor's approval.
* Other protocol inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
Phase 1b: Frequency of dose limiting toxicities (DLT) at each dose level associated with administration of copanlisib and nivolumab | At the end of Cycle 2 of a 28-day cycle
Phase 2: Overall response rate (ORR) as per RECIST v 1.1 (Response evaluation criteria in solid tumors, v 1.1) (by local investigator | Up to 26 months

SECONDARY OUTCOMES:
Phase 1b: Overall response rate (ORR) as per RECIST v 1.1 (by local investigator assessment) | Up to 26 months
Phase 1b and 2:Maximum drug concentration in plasma (Cmax) of copanlisib | At cycle1 day15, cycle2 day15, cycle 6 day15
Phase 1b and 2:Area under the curve (AUC) of copanlisib | At cycle1 day15, cycle2 day15,cycle 6 day15
Phase 1b and 2: Cmax for nivolumab | At cycle1 day15, cycle2 day15,cycle 6 day15
Phase 1b and 2: Minimum plasma drug concentration (Cmin) for nivolumab | At cycle1 day15, cycle2 day15,cycle 6 day15
Phase 1b and 2: Overall survival (OS) | Up to 26 months
Phase 1b and 2: Progression-free survival (PFS) | Up to 26 months
Phase 1b and 2: Disease control rate (DCR) | Up to 26 months
Phase 1b and 2: Duration of stable disease (DSD) | Up to 26 months
Phase 1b and 2: Time to response (TTR) | Up to 26 months
Phase 1b and 2: Time to progression (TTP) | Up to 26 months
Phase 1b and 2: Duration of response (DOR) | Up to 26 months
Phase 1b and 2:Number of participants with Adverse events (AE) and Serious AEs (SAE) | Up to 26 months
Phase 1b and 2:Number of participants with clinically significantly abnormal changes in electrocardiograms (ECG) including heart rate and measures PR, QRS, QT, and QTc intervals | Up to 26 months
Phase 1b and 2:Number of participants with changes in dose including interruptions, reductions and dose intensity | Up to 26 months

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - Tower Hematology/Oncology Medical Group, Beverly Hills, California
  - Orthopaedic Institute for Children, Los Angeles, California
  - Rocky Mountain Cancer Centers / Denver, CO, Denver, Colorado
  - Gabrail Cancer Center, Canton, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/